CLINICAL TRIAL: NCT04698746
Title: Pericapsular Nerve Group (PENG) Block Versus Intra-articular Injection for Hip Arthroscopy: A Randomized Trial
Brief Title: PENG vs Intra-articular Injection for Hip Arthroscopy
Acronym: PARİAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Serdar Yeşiltaş, Assist Prof, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 71306642-050.05.04-
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use; Acute Pain
Keywords: Hip arthroscopy, intra-articular injection, PENG block
MeSH Terms: conditions — Acute Pain | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound guided pericapsular nerve group block (Active Comparator): Injection of 15 ml 0.5% bupivacaine + 2 mg dexamethasone + 14.5 ml isotonic saline mixture between iliopubic eminentia and psoas tendon under ultrasound guidance
  Interventions: Procedure: Pericapsular nerve group block
- Intra-articular local anesthetic injection (Active Comparator): At the end of the surgical case, a total of 10 ml 0.5% bupivacaine + 2 mg dexamethasone + 9.5 ml isotonic saline injection intra-articularly.
  Interventions: Procedure: Intra-articular local anesthetic injection

INTERVENTIONS:
Procedure: Pericapsular nerve group block — PENG block will be made with 15 ml 0.5% bupivacaine + 2 mg dexamethasone + 14.5 ml NaCl under US-guidance
  Arms: Ultrasound guided pericapsular nerve group block
Procedure: Intra-articular local anesthetic injection — Intra-articular local anesthetic injection will be made with 10 ml 0.5% bupivacaine + 2 mg dexamethasone + 9.5 ml NaCl
  Arms: Intra-articular local anesthetic injection

SUMMARY:
Hip arthroscopy is a popular surgical method that is increasingly being used for both intraarticular and extraarticular hip surgeries. Postoperative acute pain is difficult to control in hip surgeries due to the complex nature of hip innervation and the large number of surgical interventions. Optimal treatment of postoperative pain in hip arthroscopy is very important to be able to perform rehabilitation, avoid opioid side effects and minimize unplanned re-hospitalization. Regional anesthesia techniques are widely used because of their proven efficacy in post-surgical pain management and their safety profile that ultimately contributes to early recovery. Many regional techniques such as neuraxial blocks, lumbar plexus block, femoral nerve block, fascia iliac block and intraarticular local anesthetic injection have been used for the treatment of acute postoperative pain.

Femoral nerve and fascia iliac blocks have shown good results for long-term post-surgery analgesia. However, the obturator nerve and accessory obturator nerve should be targeted to achieve more effective perioperative pain control. There are studies reporting that pericapsular nerve group block (PENG), which has been defined in recent years, provides effective perioperative analgesia in hip surgeries. In this study, we aim to compare the effectiveness of PENG block and intra-articular local anesthetic injection in hip arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* American Association of Anesthesiologists (ASA) physical status I - III
* BMI 20 to 35 kg / m2
* Patients scheduled for elective hip arthroscopy
* Able to provide informed consent.

Exclusion Criteria:

* Patients who refuse to participate in the study,
* Coagulopathy,
* Sepsis,
* Hepatic or renal insufficiency,
* Pregnancy
* Allergy to local anesthetic drugs,
* Chronic pain condition requiring opioid intake at home,
* BMI above 40.
* History of psychiatric diseases needing treatment.
* Failure of nerve block
* Substance abuse history
* Hip revision surgery
* Underlying neurologic disorder affecting pain perception.
* Angina, heart attack, heart failure
* Kidney or hepatic insufficiency
* Stroke
* Gastrintestinal bleeding history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | up to the first 24 hours postoperatively
  Total amount of morphine consumption during the first 24 hours after surgery. Patient controlled analgesia to be inserted.

SECONDARY OUTCOMES:
Pain intensity score | 0.5, 1, 3, 6, 12, 24 hours postoperatively.
  Postoperative pain assessed with verbal rating scale (VRS 0: no pain 10:pain as bad as can be ) at 0.5, 1, 3, 6, 12, 24 hours postoperatively.
First rescue analgesic time | up to the first 24 hours postoperatively
  The investigators will collect time to first rescue analgesic consumption in each group
Postoperative nausea and vomiting | up to the first 24 hours postoperatively
  Nausea and vomiting intensity score measured by numeric rank score (0:no nausea and no vomiting, 1: have nausea, no vomiting, 2: once vomiting, 3: two or more vomiting).
Patient satisfaction | at the end of 24 hours postoperatively
  Patient satisfaction measured using a numeric rating scale 0 to 10 (0 = unsatisfied; 10 =very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Yeşiltaş, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)